CLINICAL TRIAL: NCT04431544
Title: AcQMap® US Registry of Procedural and Long-term Clinical Outcomes (Discover-US)
Status: Terminated | Type: Observational
Why Stopped: Sponsor no longer performing clinical studies. Will only be a manufacturer
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CLP-20
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Ablation of Arrhythmia's
Keywords: ablation; atrial arrhythmia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: AcQMap System — To evaluate procedural and long-term outcomes when using the diagnostic AcQMap System as an imaging and mapping system for ablation of arrhythmias in accordance with the Instructions for Use (IFU).

SUMMARY:
AcQMap Registry is an observation study

DETAILED DESCRIPTION:
AcQMap Registry is an observational, prospective, multi-center, open-label registry designed to provide clinical data regarding the commercial, real-life experience with the diagnostic AcQMap System.

ELIGIBILITY:
Inclusion Criteria:

Male or female 18 years of age or older. Currently scheduled for an ablation of an arrhythmia utilizing the diagnostic AcQMap System.

Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study.

Willing and able to give written informed consent.

Exclusion Criteria:

In the opinion of the Investigator, any known contraindications to an ablation procedure.

Current enrollment in any study protocol sponsored by Acutus Medical. Any other condition that, in the judgment of the investigator, makes the participant a poor candidate for this procedure, the study, or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, extensive travel away from the research center, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any participant 18 years of age or older. Currently scheduled for an ablation of an arrhythmia utilizing the diagnostic AcQMap System.
Sampling Method: Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Procedural Ablation Outcomes | 12 hours
  Number of participants who had termination of ablated arrhythmia's to Sinus Rhythm or another arrhythmia within 12 hours post ablation procedure with or without electrical or pharmacological cardioversion

SECONDARY OUTCOMES:
Long-term Outcome | 3 years
  First-procedure freedom from any arrhythmia on and/or off AADs, throughout the follow-up period, excluding events in the initial 90 days following the procedure (blanking period).

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Grandview Medical Group Research, Birmingham, Alabama
  - Banner University Medical Institute, Phoenix, Arizona
  - St Jude Medical Center, Fullerton, California
  - University California San Diego, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - Mission Heritage Mission Viejo - Cardiac Electrophysiology, Mission Viejo, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Dignity Health Research Institute, Sacramento, California
  - Bethesda Hospital East, Boynton Beach, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Ascension St. Vincent's Medical Center Riverside, Jacksonville, Florida
  - Celebration Hospital, Orlando, Florida
  - Sarasota Memorial Research Institute, Sarasota, Florida
  - Bayfront (Orlando Health), St. Petersburg, Florida
  - Saint Alphonsus Health System, Boise, Idaho
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Baptist Lexington Medical Center, Lexington, Kentucky
  - Henry Ford Health Center, Detroit, Michigan
  - Nevada Heart and Vascular, Las Vegas, Nevada
  - Morristown Medical Center, Morristown, New Jersey
  - Weill Cornell Medicine, New York Presbyterian Hospital, New York, New York
  - ProMedica Physician Cardiology, Toledo, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Methodist Healthcare, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided